CLINICAL TRIAL: NCT03332810
Title: Community-based Mental Wellness Project for Adolescents and Adults: Healthy Community Pilot Project RCT Study
Brief Title: Healthy Community Pilot Project RCT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Council of Social Service (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, School of Nursing, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPH-MHP-HKCSS01
Record Dates: First submitted 2017-10-29; First posted 2017-11-06 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Mental Well-being; Happiness
Keywords: Mental health; Mental well-being; Community-based engagement; Positive psychology; Public health approach
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SME family based physical activity (Experimental): Adults and family members will participate into one core session and one booster session
  Interventions: Behavioral: SME family based physical activity
- Gathering activity (Active Comparator): Adults and family members will participate into two gathering activities
  Interventions: Behavioral: Gathering activity

INTERVENTIONS:
Behavioral: SME family based physical activity — * One train-the-trainer workshop: to train the service providers from 8-15 NGO service units on the concept of SME, ways of conducting mental well-being activities and knowledge of adult mental health problem (in particular the mixed anxiety and depressive disorder).
  * Two SME family-based physical activities held by each NGO service unit: to organize enjoyable activities according to the needs of individual district as well as to promote positive psychology under the theme of SME. All these activities are organized by the NGO service providers in collaboration with District Healthy City Committee.
  Arms: SME family based physical activity
Behavioral: Gathering activity — - Gathering activities will be held for control groups. However, SME concept or techniques will not be introduced during the activity. Physical activity will not be used as the intervention method.
  Arms: Gathering activity

SUMMARY:
Aims: To enhance mental well-being of adolescents, adults and their families by creating a positive, happy and joyful environment in the community.

Targets: Adults aged 18-59 and their family members in Hong Kong.

Methods: Healthy Community Pilot Project will adopt the public health and family-focused approach, under the brand name of "Joyful@HK Campaign". Evidence-based and Evidence Generating approach with vigorous study design, both qualitative (e.g. focus groups) and quantitative (e.g. randomised controlled trial), will be used to evaluate the overall programme effectiveness including follow-up of at least one month ("best science"). To ensure the practicability and sustainability of the community-based engagement project, we will engage community partners with strong track records of "best practice" to design, plan, and implement the intervention. This project will use innovative and integrated positive psychology and public health theories and methods to plan brief, simple, and cost-effective intervention.

Significance: By using "best science" in the design and evaluation of intervention programme, and the "best practice" of the partners' skills, experience and strong connection with service targets in the community, the intervention, if proven to be effective, for promoting sharing, mind and enjoyment and enhancing mental well-being can be further developed and widely disseminated to and adopted by the practitioners in the health and social service sectors for replication and improvement to benefit the whole population.

DETAILED DESCRIPTION:
Healthy Community Pilot Project is one of the six Community-based Mental Wellness Project for Adolescents and Adults, which aims at enhancing mental well-being of adolescents, adults and their families by creating a positive, happy and joyful environment in the community. The project is funded by Health Care and Promotion Fund of Food and Health Bureau.

Healthy Community Pilot Project is organized by the Hong Kong Council of Social Service and led by the School of Public Health, The University of Hong Kong.The project will organize one train-the-trainer workshop to train the service providers from 8-10 NGO service units on the concept of sharing, mind and enjoyment (SME), ways of conducting SME family-based physical activities and knowledge of adult mental health problem (in particular the mixed anxiety and depressive disorder). Two SME family-based physical activities will be held by the NGO service providers in collaboration with 3 District Healthy City Committees. Each NGO service unit may organize enjoyable SME family-based physical activities according to the needs of individual district and to promote positive psychology under the theme of Sharing, Mind and Enjoyment. One wisdom sharing session will be organized to members of District Healthy City Committees to promote best practice of community mental wellness project.

The major subjects of the Healthy Community Pilot Project RCT study are 150-200 families with 400 participants. 3 District Healthy City Committees will be selected as collaborators. 10-18 NGO service units will either be randomized into intervention service units and control service units. Cluster Randomized Control Trial will be used to evaluate the effectiveness of the intervention programme.

In the study, families will be invited to complete a series of questionnaires or invited to attend focus groups to measure the sharing, mind and enjoyment related behavioural changes, mental well-being and subjective changes. NGO workers who joined the train-the-trainer workshop will also be invited to complete questionnaires to measure their knowledge about mental health, skills of conducting SME family-based physical activities and their sharing, mind and enjoyment related behavioural change. They will be invited to focus group interview to assess their experience and feedback on this project while community partners will be invited to individual in-depth interviews to assess the outcomes of community engagement process.

HKU team will conduct evaluation during the programme implementation stage. The effectiveness of the intervention, as well as the level of participation and ratings for the intervention will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Families (Major subjects):

   * Adults aged 18-59 and their family members (Their family members could be children)
   * Chinese speaking
   * Able to complete study questionnaires/ focus groups
2. Service providers of NGO service units

   * Staff working in the participating NGO service units
   * Adults aged 18-59
   * Chinese speaking
   * Able to complete study questionnaires/ focus group
3. Community partners

   * Staff working in the collaborating NGO service units or District Healthy City Committees in partnership with HKU research team to organize or plan or implement the project
   * Chinese speaking
   * Able to complete study questionnaires/ individual in-depth interviews

Exclusion Criteria:

* Those who cannot read Chinese
* Those who suffered from severe mental disorders

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in participants' frequency of performing the suggested Sharing, Mind and Enjoyment (SME) related behaviours | T1: baseline; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  The frequency of performing the SME (Sharing: encourage families to do physical activity, encourage families to do zero-time exercise, do physical activity with families; Mind: have intention, goal and confidence to do physical activity; Enjoyment: enjoy physical activity) related behaviours in the past 7 days will be assessed. The questions are rated 0-7 with 0 indicating none of this behavior happened in the past 7 days and 7 indicating this behavior happened every day in the past 7 days.

SECONDARY OUTCOMES:
Changes in personal happiness from baseline to three-month after baseline | T1: baseline; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  Personal happiness will be assessed by Subjective Happiness Scale (SHS). SHS was rated on 7-point scale with 1 indicating not happiness at all and 7 indicating extreme happiness. To score the scale, the 4th item will be coded reversely and mean of the 4 items will be computed.
Changes in mental well-being from baseline to three-month after baseline | T1: baseline; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  Mental well-being will be assessed by validated Chinese version of 7-item Warwick Edinburgh Well-being Scale. Each item ranges from 1 to 5 and the scale will be scored by first summing the score for each of the 7 items and then transforming the total score for each person according to a conversion table.
Changes in family relationship from baseline to three-month after baseline | T1: baseline; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  Self-perceived understanding, intimacy, and family communication will be assessed by three questions (rated 0-10).
Changes in individual and family health from baseline to three-month after baseline | T1: baseline; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  Self-perceived health, at the individual and family level will be assessed by two questions respectively (rated 0-10).
Changes in individual and family happiness from baseline to three-month after baseline | T1: baseline; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  Self-perceived happiness, at the individual and family level will be assessed by two questions respectively (rated 0-10).
Changes in family harmony from baseline to three-month after baseline | T1: baseline; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  Self-perceived family harmony will be assessed by a single question (rated 0-10).
Changes in knowledge and perception of mixed anxiety and depressive disorders | T1: baseline; T2: immediate post intervention; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  Knowledge and perception of mixed anxiety and depressive disorders will be assessed by 4 questions (2 questions about understanding of symptoms, 1 about the intention of help seeking, 1 about support seeking from families) rated 0-10.
Satisfaction towards SME physical activity training & program | T2: immediate post intervention; T3: one-month follow-up after baseline
  Satisfaction towards programme will be assessed by conducting focus group and program evaluation measures (general satisfaction, self-perceived helpfulness and likely-to-recommend level) rated 0-10.
The social impact of the community-based engagement project | Up to four months
  The social impact of the community-based engagement project will be evaluated by conducting community stakeholders' in-depth interviews.
The process of community based intervention programme | Up to four months
  Assessed by a Process Evaluation on-site observation form, and a series of checklists including Resources input record sheet, Participants' attendance form, Programme rundown, Attendance record form, and NGOs' final report. The components of process evaluation, including context, reach, dose delivered, dose received, fidelity and recruitment will be assessed.
Outcomes of community engagement process | Up to four months
  Outcomes of community engagement process will be assessed by a self-designed questionnaire survey.

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, Principal Investigator — The University of Hong Kong
Locations (1):
- The Hong Kong Council of Social Service, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun Y, Ho SY, Chan CS, Wang MP, Wan ANT, Xu Y, Lai AYK, Lam TH. Brief Intervention to Promote Physical Activity and Mental Well-Being in Community Adults: A Pilot Cluster Randomized Controlled Trial. J Prim Care Community Health. 2024 Jan-Dec;15:21501319241281567. doi: 10.1177/21501319241281567. PMID 39279371